CLINICAL TRIAL: NCT04806165
Title: Developing an Optimized Conversational Agent or "Chatbot" to Facilitate Mental Health Services Use in Individuals With Eating Disorders
Brief Title: Treatment Uptake Chatbot for Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 202007008; K08MH120341 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Repeated Administration (Experimental)
  Interventions: Behavioral: Repeated Administration
- Personalized Recommendation (Experimental)
  Interventions: Behavioral: Personalized Recommendation
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Core Modules Only (Experimental)
  Interventions: Behavioral: Core Modules Only
- Motivational Interviewing, Personalized Recommendation, Repeated Administration (Experimental)
  Interventions: Behavioral: Motivational Interviewing, Personalized Recommendation, Repeated Administration
- Motivational Interviewing, Repeated Administration (Experimental)
  Interventions: Behavioral: Motivational Interviewing, Repeated Administration
- Motivational Interviewing, Personalized Recommendation (Experimental)
  Interventions: Behavioral: Motivational Interviewing, Personalized Recommendation
- Personalized Recommendation, Repeated Administration (Experimental)
  Interventions: Behavioral: Personalized Recommendation, Repeated Administration
- Psychoeducation (Experimental)
  Interventions: Behavioral: Psychoeducation
- Psychoeducation, Repeated Administration (Experimental)
  Interventions: Behavioral: Psychoeducation, Repeated Administration
- Psychoeducation, Personalized Recommendation (Experimental)
  Interventions: Behavioral: Psychoeducation, Personalized Recommendation
- Psychoeducation, Motivational Interviewing (Experimental)
  Interventions: Behavioral: Psychoeducation, Motivational Interviewing
- Psychoeducation, Motivational Interviewing, Personalized Recommendation (Experimental)
  Interventions: Behavioral: Psychoeducation, Motivational Interviewing, Personalized Recommendation
- Psychoeducation, Personalized Recommendation, Repeated Administration (Experimental)
  Interventions: Behavioral: Psychoeducation, Personalized Recommendation, Repeated Administration
- Psychoeducation, Motivational Interviewing, Repeated Administration (Experimental)
  Interventions: Behavioral: Psychoeducation, Motivational Interviewing, Repeated Administration
- Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration (Experimental)
  Interventions: Behavioral: Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration

INTERVENTIONS:
Behavioral: Repeated Administration — A discussion with the chatbot, including follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Repeated Administration
Behavioral: Personalized Recommendation — A discussion with the chatbot, including identifying a personalized recommendation for accessing help for their eating disorder.
  Arms: Personalized Recommendation
Behavioral: Motivational Interviewing — A discussion with the chatbot, including motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder.
  Arms: Motivational Interviewing
Behavioral: Core Modules Only — A discussion with the chatbot, including only the core modules.
  Arms: Core Modules Only
Behavioral: Motivational Interviewing, Personalized Recommendation, Repeated Administration — A discussion with the chatbot, including motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder, identifying a personalized recommendation for accessing help for their eating disorder, and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Motivational Interviewing, Personalized Recommendation, Repeated Administration
Behavioral: Motivational Interviewing, Repeated Administration — A discussion with the chatbot, including motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Motivational Interviewing, Repeated Administration
Behavioral: Motivational Interviewing, Personalized Recommendation — A discussion with the chatbot, including motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder and identifying a personalized recommendation for accessing help for their eating disorder.
  Arms: Motivational Interviewing, Personalized Recommendation
Behavioral: Personalized Recommendation, Repeated Administration — A discussion with the chatbot, including identifying a personalized recommendation for accessing help for their eating disorder and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Personalized Recommendation, Repeated Administration
Behavioral: Psychoeducation — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders.
  Arms: Psychoeducation
Behavioral: Psychoeducation, Repeated Administration — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Psychoeducation, Repeated Administration
Behavioral: Psychoeducation, Personalized Recommendation — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders and identifying a personalized recommendation for accessing help for their eating disorder.
  Arms: Psychoeducation, Personalized Recommendation
Behavioral: Psychoeducation, Motivational Interviewing — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders and motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder.
  Arms: Psychoeducation, Motivational Interviewing
Behavioral: Psychoeducation, Motivational Interviewing, Personalized Recommendation — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders, motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder, and identifying a personalized recommendation for accessing help for their eating disorder.
  Arms: Psychoeducation, Motivational Interviewing, Personalized Recommendation
Behavioral: Psychoeducation, Personalized Recommendation, Repeated Administration — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders, identifying a personalized recommendation for accessing help for their eating disorder, and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Psychoeducation, Personalized Recommendation, Repeated Administration
Behavioral: Psychoeducation, Motivational Interviewing, Repeated Administration — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders, motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder, and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Psychoeducation, Motivational Interviewing, Repeated Administration
Behavioral: Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration — A discussion with the chatbot, including psychoeducational content to increase knowledge related to eating disorders, motivational interviewing techniques to help overcome barriers to seeking care for their eating disorder, identifying a personalized recommendation for accessing help for their eating disorder, and follow ups over the course of 2 weeks to encourage help seeking for their eating disorder.
  Arms: Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration

SUMMARY:
Eating disorders (EDs) are serious mental illnesses associated with high morbidity and mortality, clinical impairment, and comorbid psychopathology. Although evidence-based treatments for EDs have been established, the treatment gap is wide. Indeed, <20% of individuals with EDs receive treatment. There is need for a novel solution not only to identify individuals with EDs but also to encourage mental health services use and to address treatment barriers. This study aims to implement a conversational agent or "chatbot" that is optimized to increase mental health services use among individuals with EDs through such features as: 1) education on the seriousness and consequences of EDs; 2) engaging the user in motivational interviewing to overcome barriers to care; 3) providing a personalized recommendation for seeking intervention; 4) repeated check-ins with the user to encourage follow-up with care. This study will utilize a randomized optimization trial with adults who have completed screening on the National Eating Disorders Association (NEDA) website and screen positive for an ED but are not in treatment to determine chatbot feasibility and to generate data on the effect of the chatbot on motivation for treatment and mental health services use. This trial will employ the Multiphase Optimization Strategy framework, using a 2^4 full factorial design, to randomly assign participants to a combination of the four proposed intervention components (n=16 conditions) to isolate the active ingredients.

ELIGIBILITY:
Inclusion Criteria:

* U.S. resident
* English-speaking
* Age 18 years or older
* Owns a personal smartphone
* Screens positive for a Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) clinical or subclinical eating disorder
* Not currently receiving treatment for an eating disorder

Exclusion Criteria:

* Non-U.S. resident
* Younger than 18 years old
* Does not own a personal smartphone
* Does not screen positive for a DSM-5 clinical or subclinical eating disorder
* Screens positive for Avoidant Restrictive Food Intake Disorder
* Currently receiving treatment for an eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Fitzsimmons-Craft, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who completed the NEDA screen and met all eligibility criteria were shown the baseline assessment. Individuals who completed the baseline, were U.S. residents, and endorsed owning a smartphone were shown the consent form. N= 205 individuals provided consent and were randomized to a condition.
Period: Overall Study
Arm/Group | Repeated Administration | Personalized Recommendation | Motivational Interviewing | Core Modules Only | Motivational Interviewing, Personalized Recommendation, Repeated Administration | Motivational Interviewing, Repeated Administration | Motivational Interviewing, Personalized Recommendation | Personalized Recommendation, Repeated Administration | Psychoeducation | Psychoeducation, Repeated Administration | Psychoeducation, Personalized Recommendation | Psychoeducation, Motivational Interviewing | Psychoeducation, Motivational Interviewing, Personalized Recommendation | Psychoeducation, Personalized Recommendation, Repeated Administration | Psychoeducation, Motivational Interviewing, Repeated Administration | Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration
Started | 13 | 12 | 11 | 14 | 13 | 13 | 14 | 13 | 13 | 12 | 13 | 13 | 13 | 13 | 12 | 13
Completed 2-Week Follow-Up Assessment | 10 | 9 | 10 | 12 | 11 | 8 | 10 | 9 | 10 | 10 | 10 | 8 | 10 | 9 | 9 | 11
Completed 6-Week Follow-Up Assessment | 9 | 8 | 9 | 10 | 9 | 7 | 8 | 9 | 9 | 11 | 9 | 8 | 10 | 9 | 9 | 10
Completed 14-Week Follow-Up Assessment | 9 | 10 | 9 | 10 | 10 | 6 | 10 | 9 | 9 | 11 | 10 | 8 | 9 | 8 | 6 | 11
Completed | 13 | 12 | 11 | 14 | 13 | 13 | 14 | 13 | 13 | 12 | 13 | 13 | 13 | 13 | 12 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Following screening, individuals were shown the baseline assessment link if they met the following eligibility criteria: screened positive for a clinical/subclinical ED, not currently in treatment for an ED, and at least 18 years old. U.S residents who completed the baseline assessment and endorsed owning a smartphone were offered to participate and shown the consent form. N=205 individuals provided sent and were randomized to one of sixteen conditions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Repeated Administration | Personalized Recommendation | Motivational Interviewing | Core Modules Only | Motivational Interviewing, Personalized Recommendation, Repeated Administration | Motivational Interviewing, Repeated Administration | Motivational Interviewing, Personalized Recommendation | Personalized Recommendation, Repeated Administration | Psychoeducation | Psychoeducation, Repeated Administration | Psychoeducation, Personalized Recommendation | Psychoeducation, Motivational Interviewing | Psychoeducation, Motivational Interviewing, Personalized Recommendation | Psychoeducation, Personalized Recommendation, Repeated Administration | Psychoeducation, Motivational Interviewing, Repeated Administration | Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration | Total
Number analyzed (Participants) | 13 | 12 | 11 | 14 | 13 | 13 | 14 | 13 | 13 | 12 | 13 | 13 | 13 | 13 | 12 | 13 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.31 (7.71) | 29.50 (8.19) | 36.27 (13.98) | 38.42 (15.32) | 30.69 (10.93) | 37.69 (14.85) | 29.57 (7.74) | 29.57 (7.74) | 40.46 (18.33) | 29.15 (9.51) | 32.42 (13.34) | 39.31 (14.06) | 31.10 (10.65) | 30.38 (12.47) | 32.38 (13.12) | 34.58 (14.09) | 30.00 (9.41)
Age, Customized [Number; unit: participants]
  18-24 | 6 | 2 | 2 | 3 | 5 | 3 | 3 | 4 | 5 | 3 | 2 | 4 | 6 | 4 | 4 | 5 | 61
  25-34 | 5 | 7 | 4 | 4 | 4 | 3 | 9 | 2 | 5 | 4 | 3 | 5 | 3 | 5 | 3 | 5 | 71
  35-44 | 1 | 3 | 2 | 1 | 2 | 2 | 1 | 1 | 2 | 3 | 4 | 1 | 1 | 2 | 3 | 2 | 31
  45-54 | 1 | 0 | 2 | 3 | 2 | 4 | 1 | 3 | 1 | 0 | 2 | 3 | 3 | 1 | 1 | 0 | 27
  55-64 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 11
  65-74 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 14 | 11 | 12 | 13 | 13 | 11 | 11 | 13 | 11 | 13 | 10 | 10 | 13 | 184
  Male | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 12
  Non-binary/third gender | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 7
  Prefer not to say | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 9 | 10 | 10 | 14 | 12 | 13 | 14 | 13 | 12 | 11 | 13 | 13 | 13 | 11 | 11 | 13 | 192
    Male | 4 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 17
  Not Hispanic or Latino | 12 | 11 | 10 | 14 | 12 | 10 | 13 | 12 | 12 | 12 | 13 | 11 | 11 | 12 | 11 | 12 | 188
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 0 | 0 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  White | 11 | 9 | 9 | 12 | 11 | 9 | 11 | 9 | 12 | 12 | 11 | 9 | 9 | 11 | 10 | 8 | 163
  More than one race | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 16
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 11 | 14 | 13 | 13 | 14 | 13 | 13 | 12 | 13 | 13 | 13 | 13 | 12 | 13 | 205

OUTCOME MEASURES:

1. Primary Outcome: Rates of Treatment/Services Utilization for Eating, Shape, or Weight Concerns Among All Participants Randomized to the Intervention Following Online Eating Disorder Screening
Description: Treatment utilization was measured at each follow-up time point (2, 6, and 14 weeks), which was assessed via the prompt, "Have you tried or used any type of mental health help (e.g., self-help app, telehealth/in-person counseling, etc.) for your concerns related to your eating, shape, or weight in the past [2, 6, or 14] weeks?". We defined a participant as having utilized treatment at the first time they responded, "yes" (vs. "no") to this question. The data presented below indicate the rates of self-reported receipt of treatment/services utilization among participants assigned (component on) or not assigned (component off) to each of the four chatbot components (motivational interviewing, psychoeducation, personalized recommendations, repeated administration), as delineated by each time point during which the aforementioned item was assesed.
Time Frame: 2, 6, 14 Weeks from Engagement with the Intervention
Population: All participants who engaged with the intervention and completed the treatment utilization item at each follow up assessment (2, 6, and 14 weeks post intervention) are included. Participants in each of the 16 factorial conditions were sorted based on whether or not each of the four chatbot components were assigned. This method was used in order to understand which combination of components are essential in the design of an optimized chatbot for use in a future randomized controlled trial.
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interviewing On: Participants were randomized to a chatbot condition that included the motivational interviewing component of the conversation (i.e., the motivational interviewing component was turned on during the chatbot conversations of these participants).
- Motivational Interviewing Off: Participants were randomized to a chatbot condition that did not include the motivational interviewing component of the conversation (i.e., the motivational interviewing component was turned off during the chatbot conversations of these participants).
- Personalized Recommendation On: Participants were randomized to a chatbot condition that included the personalized recommendations component of the conversation (i.e., the personalized recommendations component was turned on during the chatbot conversations of these participants).
- Personalized Recommendation Off: Participants were randomized to a chatbot condition that did not include the personalized recommendations component of the conversation (i.e., the personalized recommendations component was turned off during the chatbot conversations of these participants). Instead, these participants received general recommendations for treatment and services.
- Psychoeducation On: Participants were randomized to a chatbot condition that included the psychoeducation component of the conversation (i.e., the psychoeducation component was turned on during the chatbot conversations of these participants).
- Psychoeducation Off: Participants were randomized to a chatbot condition that did not include the psychoeducation component of the conversation (i.e., the psychoeducation component was turned off during the chatbot conversations of these participants).
- Repeated Administration On: Participants were randomized to a chatbot condition that included the repeated administration component of the conversation (i.e., the repeated administration component was turned on during the chatbot conversations of these participants). Participants in this group received up to three check-ins from the chatbot over the course of the next 9 days. At the first check-in, which occurred 3 days after the main conversation, the chatbot asked users if they had sought help or used any of the recommended tools/services since they last conversed. If users do not report seeking help and/or utilizing services, they continued to receive check-ins until treatment receipt was provided.
- Repeated Administration Off: Participants were randomized to a chatbot condition that did not include the repeated administration component of the conversation (i.e., the repeated administration component was turned off during the chatbot conversations of these participants). Participants in this group completed the main conversation with the chatbot, which consisted of the introduction, a combination of the motivational interviewing, personalized recommendation, and psychoeducation components (which was determined by which of the 16 conditions participants were randomized to), and the corresponding conclusion. The conversation with the chatbot terminated following the conclusion, and the chatbot did not message users subsequently (unless users reached out to the chatbot first).
Arm/Group | Motivational Interviewing On | Motivational Interviewing Off | Personalized Recommendation On | Personalized Recommendation Off | Psychoeducation On | Psychoeducation Off | Repeated Administration On | Repeated Administration Off
Number analyzed (Participants) | 67 | 74 | 73 | 68 | 70 | 71 | 71 | 70
Participants
  Number of Participants Reporting New Treatment Receipt at 2 Weeks from Baseline | 40 | 41 | 45 | 36 | 42 | 39 | 46 | 35
  Number of Participants Reporting New Treatment Receipt at 6 Weeks from Baseline: number analyzed (Participants) | 27 | 33 | 28 | 32 | 28 | 32 | 25 | 35
  Number of Participants Reporting New Treatment Receipt at 6 Weeks from Baseline | 5 | 10 | 8 | 7 | 3 | 12 | 5 | 10
  Number of Participants Reporting New Treatment Receipt at 14 Weeks from Baseline: number analyzed (Participants) | 22 | 23 | 20 | 25 | 25 | 20 | 20 | 25
  Number of Participants Reporting New Treatment Receipt at 14 Weeks from Baseline | 6 | 9 | 6 | 9 | 8 | 7 | 8 | 7
  Cumulative Sum of Participants Reporting Treatment Receipt over Study Period | 51 | 60 | 45 | 36 | 42 | 39 | 46 | 35
Statistical Analysis 1: Comparison: Motivational Interviewing On vs Motivational Interviewing Off; This analysis explores the effect of the motivational interviewing (MI) component on rates of treatment receipt over the entire study period. Results will help determine the proportional increase in odds of treatment seeking corresponding to receiving each chatbot component. Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — To improve the quality of the imputations, gender, age, and race were included as auxiliary variables. We generated ten imputed datasets with the predictive mean matching method and pooled coefficients, degrees of freedom, and standard errors with Rubin's (1987) rules. As a sensitivity analysis, we also ran the same models using full information maximum likelihood to handle missing data. The model was estimated using a logit link and did not incorporate an intercept; p = .309, Discrete Time Survival Analysis — We defined sufficiently large main effects as those with p values ≤ .05 or with 95% confidence intervals that do not include 0. We interpreted absolute ß values below 0.2 as small, between 0.2 and 0.5 as medium, and greater than 0.5 as large; The model did not incorporate an intercept to allow for estimation of treatment receipt likelihood among participants yet to report treatment; Regression (Beta) Coefficient = -.26, Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Personalized Recommendation On vs Personalized Recommendation Off; This analysis explores the effect of the personalized recommendation (PR) component on rates of treatment receipt over the entire study period. Results will help determine the proportional increase in odds of treatment seeking corresponding to receiving each chatbot component. Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .190, Discrete Time Survival Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Regression (Beta) Coefficient = .34, Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Psychoeducation On vs Psychoeducation Off; This analysis explores the effect of the psychoeducation (PE) component on rates of treatment receipt over the entire study period. Results will help determine the proportional increase in odds of treatment seeking corresponding to receiving each chatbot component. Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .690, Discrete Time Survival Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Regression (Beta) Coefficient = -0.10, Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Repeated Administration On vs Repeated Administration Off; This analysis explores the effect of the repeated administration (RA) component on rates of treatment receipt over the entire study period. Results will help determine the proportional increase in odds of treatment seeking corresponding to receiving each chatbot component. Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.038, Discrete Time Survival Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Regression (Beta) Coefficient = 0.54, Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis provides results on the 2 week time point post Intervention and contributes to understanding of the effect of time since chatbot engagement on treatment receipt, regardless of the combination of the four chatbot components participants were assigned (ie., component turned off or on). Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .735, Discrete Time Survival Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Regression (Beta) Coefficient = 0.06, Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis provides results on the 6 week time point post Intervention and contributes to understanding of the effect of time since chatbot engagement on treatment receipt, regardless of the combination of the four chatbot components participants were assigned (ie., component turned off or on). Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .001, Discrete Time Survival Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Regression (Beta) Coefficient = -0.91, Standard Error of Mean 0.27
Statistical Analysis 7: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis provides results on the 14 week time point post Intervention and contributes to understanding of the effect of time since chatbot engagement on treatment receipt, regardless of the combination of the four chatbot components participants were assigned (ie., component turned off or on). Discrete time survival analysis was employed and models were fit with treatment seeking regressed on follow-up time (2-week, 6-week, or 14-week) and each chatbot component; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = .014, Discrete Time Survival Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Regression (Beta) Coefficient = -0.73, Standard Error of Mean 0.30

2. Secondary Outcome: Mean Willingness to Seek Psychotherapy
Description: Participants' willingness to seek psychotherapy was assessed via an identical item in the baseline assessment (i.e., before the initial chatbot assessment) as well as each off the follow-up assessments delivered at 2, 6, and 14 weeks post-intervention. The item prompted users to rate their willingness to seek in-person or telehealth psychotherapy in subsequent weeks. Responses were rated on a Likert scale from 1 (not at all important/ready) to 7 (very important/ready). Mean values reported below indicate the average Likert scale willingness rating among all participants at each time point who did (component turned on) and did not (component turned off). Statistical analyses outline the time and component effects on changes in mean willingness to seek pyschotherapy from baseline to 14 weeks post-interventioon.
Time Frame: Baseline, 2 Weeks, 6 Weeks, 14 Weeks
Population: The analysis population included those individuals who did not report utilizing treatment/services at any of the three follow-up assessments. Treatment utilization was assessed via the item,"Have you tried or used any type of mental health help (e.g., self-help app, telehealth/in-person counseling, etc.) for your concerns related to your eating, shape, or weight in the past past [2, 6, or 14] weeks?" Participants who did not respond "yes" to this item were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing On | Motivational Interviewing Off | Personalized Recommendation On | Personalized Recommendation Off | Psychoeducation On | Psychoeducation Off | Repeated Administration On | Repeated Administration Off
Number analyzed (Participants) | 47 | 40 | 40 | 47 | 44 | 43 | 39 | 48
score on a scale
  Baseline | 4.64 (1.92) | 4.23 (2.03) | 4.30 (1.88) | 4.57 (2.05) | 4.30 (2.08) | 4.60 (1.87) | 4.69 (2.03) | 4.25 (1.92)
  2 Weeks from Baseline: number analyzed (Participants) | 26 | 19 | 20 | 25 | 24 | 21 | 17 | 28
  2 Weeks from Baseline | 3.88 (2.03) | 3.47 (1.90) | 3.85 (1.84) | 3.60 (2.08) | 3.96 (1.88) | 3.43 (2.06) | 4.71 (1.79) | 3.11 (1.83)
  6 Weeks from Baseline: number analyzed (Participants) | 22 | 16 | 16 | 22 | 22 | 16 | 15 | 23
  6 Weeks from Baseline | 3.77 (2.07) | 3.56 (2.13) | 4.00 (2.10) | 3.45 (2.06) | 3.86 (2.19) | 3.44 (1.93) | 3.93 (2.12) | 3.52 (2.06)
  14 Weeks from Baseline: number analyzed (Participants) | 21 | 17 | 18 | 20 | 21 | 17 | 13 | 25
  14 Weeks from Baseline | 3.71 (1.98) | 3.41 (1.77) | 3.11 (1.78) | 4.00 (1.89) | 3.62 (2.11) | 3.53 (1.59) | 3.85 (1.72) | 3.44 (1.96)
Statistical Analysis 1: Comparison: Motivational Interviewing On vs Motivational Interviewing Off; Analyses were conducted to determine the effects of each of the four chatbot components on secondary outcomes. This analysis in particular explores the effects of the motivational interviewing component (MI) on participant willingness to seek psychotherapy for concerns their disordered weight and shape behaviors and thoughts since engagement with the intervention. Linear mixed effects models incorporated a random intercept to accommodate the correlation of repeated measures within participants; Test type: Superiority — Gender, age, and race were included as auxiliary variables to improve imputation quality. We generated ten imputed datasets with the predictive mean matching method and pooled coefficients, degrees of freedom, and standard errors with Rubin's (1987) rules. For sensitivity analysis, models were run again using full information maximum likelihood to handle missing data; p = 0.25, Linear Mixed Effects Model — We interpreted absolute ß values below 0.2 as small, between 0.2 and 0.5 as medium, and greater than 0.5 as large. We defined sufficiently large main effects as those with p values ≤ .05 or with 95% confidence intervals that do not include 0; Regression (Beta) Coefficient = 0.53
Statistical Analysis 2: Comparison: Psychoeducation On vs Psychoeducation Off; Analyses were conducted to determine the effects of each of the four chatbot components on willingness to seek psychotherapy. This analysis in particular explores the effects of the psychoeducation component (PE) on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — To improve the quality of the imputations, gender, age, and race were included as auxiliary variables. We generated ten imputed datasets with the predictive mean matching method and pooled coefficients, degrees of freedom, and standard errors with Rubin's (1987) rules. As a sensitivity analysis, we also ran the same models using full information maximum likelihood to handle missing data; p = 0.44, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; The linear mixed effects models incorporated a random intercept to accommodate the correlation of repeated measures within participants; Regression (Beta) Coefficient = -0.36
Statistical Analysis 3: Comparison: Personalized Recommendation On vs Personalized Recommendation Off; Analyses were conducted to determine the effects of each of the four chatbot components on willingness to seek psychotherapy. This analysis in particular explores the effects of the personalized recommendation component (PR) on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.44, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.25
Statistical Analysis 4: Comparison: Repeated Administration On vs Repeated Administration Off; Analyses were conducted to determine the effects of each of the four chatbot components on willingness to seek psychotherapy. This analysis in particular explores the effects of the repeated administration component (RA) on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.53, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 0.29
Statistical Analysis 5: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis provides results on the 2 week time point post Intervention and contributes to understanding of the effect of time since chatbot engagement on willingness to seek psychotherapy, regardless of the combination of the four chatbot components participants were assigned (ie., component turned off or on); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.07, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.53
Statistical Analysis 6: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis provides results on the 6 week time point post Intervention and contributes to understanding of the effect of time since chatbot engagement on willingness to seek psychotherapy, regardless of the combination of the four chatbot components participants were assigned (ie., component turned off or on); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.01, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -1.06
Statistical Analysis 7: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis provides results on the 14 week time point post Intervention and contributes to understanding of the effect of time since chatbot engagement on willingness to seek psychotherapy, regardless of the combination of the four chatbot components participants were assigned (ie., component turned off or on); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.042, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.85
Statistical Analysis 8: Comparison: Motivational Interviewing On vs Motivational Interviewing Off; This analysis explores the interaction effects of 2-week time since engagement with the intervention and the motivational interviewing (MI) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.89, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.08
Statistical Analysis 9: Comparison: Motivational Interviewing On vs Motivational Interviewing Off; This analysis explores the interaction effects of 6-week time since engagement with the intervention and the motivational interviewing (MI) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.69, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 0.34
Statistical Analysis 10: Comparison: Motivational Interviewing On vs Motivational Interviewing Off; This analysis explores the interaction effects of 14-week time since engagement with the intervention and the motivational interviewing (MI) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.40, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.69
Statistical Analysis 11: Comparison: Psychoeducation On vs Psychoeducation Off; This analysis explores the interaction effects of 2-week time since engagement with the intervention and the psychoeducation (PE) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.55, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 0.35
Statistical Analysis 12: Comparison: Psychoeducation On vs Psychoeducation Off; This analysis explores the interaction effects of 6-week time since engagement with the intervention and the psychoeducation (PE) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.32, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 0.88
Statistical Analysis 13: Comparison: Psychoeducation On vs Psychoeducation Off; This analysis explores the interaction effects of 14-week time since engagement with the intervention and the psychoeducation (PE) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.63, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.37
Statistical Analysis 14: Comparison: Personalized Recommendation On vs Personalized Recommendation Off; This analysis explores the interaction effects of 2-week time since engagement with the intervention and the personalized recommendation (PR) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.90, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 0.08
Statistical Analysis 15: Comparison: Personalized Recommendation On vs Personalized Recommendation Off; This analysis explores the interaction effects of 6-week time since engagement with the intervention and the personalized recommendation (PR) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.27, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.95
Statistical Analysis 16: Comparison: Personalized Recommendation On vs Personalized Recommendation Off; This analysis explores the interaction effects of 14-week time since engagement with the intervention and the personalized recommendation (PR) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.42, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.67
Statistical Analysis 17: Comparison: Repeated Administration On vs Repeated Administration Off; This analysis explores the interaction effects of 2-week time since engagement with the intervention and the repeated administration (RA) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.04, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 1.23
Statistical Analysis 18: Comparison: Repeated Administration On vs Repeated Administration Off; This analysis explores the interaction effects of 6-week time since engagement with the intervention and the repeated administration (RA) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.16, Multilevel Models — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 1.22
Statistical Analysis 19: Comparison: Repeated Administration On vs Repeated Administration Off; This analysis explores the interaction effects of 14-week time since engagement with the intervention and the repeated administration (RA) component on participant willingness to seek psychotherapy for concerns related to their eating, weight, and/or shape concerns. since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.99, Linear Mixed Effects Model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = 0.01

3. Secondary Outcome: Mean Attitude Toward Change for Concerns Related to Eating, Shape, or Weight Concerns Among All Participants Randomized to the Intervention Following Online Eating Disorder Screening
Description: Participants' attitudes toward making changes (i.e., motivation toward seeking help) to address their personal eating, shape, and weight concerns were measured via identical items in the baseline assessment, and in each of the 2, 6, and 14 week follow-up assessments. Items included, "How important is it for you to change your eating, shape, or weight concerns?" and, "How ready are you to make changes in your eating, shape, or weight concerns?". Both items were rated on a Likert scale from 1 (not at all important/ready) to 7 (very important/ready), and the sum of the two questions was used as an index of change/motivation attitudes. Values below indicate the average Likert scale attitude rating (from 2 (lowest) to 14 (highest)) among all participants at each time point who did (component turned on) and did not (component turned off) receive each component. Analyses outline the time, component, and time by component interaction effects on changes in motivation attitudes since baseline.
Time Frame: Baseline, 2 weeks, 6 weeks, 14 weeks
Population: All participants randomized to the intervention (n=205) were included, with missing data accommodated using maximum likelihood estimation. This study uses a factorial design; participants were randomized to one of 16 conditions, with each condition receiving a different combination of the four chatbot components (motivational interviewing, psychoeducation, personalized recommendations, repeated administration) turned off or on. Data below are presented as such.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing On | Motivational Interviewing Off | Personalized Recommendation On | Personalized Recommendation Off | Psychoeducation On | Psychoeducation Off | Repeated Administration On | Repeated Administration Off
Number analyzed (Participants) | 102 | 103 | 104 | 101 | 102 | 103 | 102 | 103
score on a scale
  Baseline: number analyzed (Participants) | 47 | 103 | 104 | 101 | 102 | 103 | 102 | 103
  Baseline | 11.80 (2.35) | 11.05 (2.89) | 11.40 (2.66) | 11.45 (2.68) | 11.40 (2.70) | 11.45 (2.63) | 11.34 (2.76) | 11.50 (2.57)
  2 Weeks from Baseline: number analyzed (Participants) | 26 | 79 | 79 | 77 | 77 | 79 | 77 | 79
  2 Weeks from Baseline | 10.73 (2.59) | 10.70 (2.95) | 10.53 (2.65) | 10.90 (2.89) | 10.31 (2.93) | 11.10 (2.57) | 10.86 (2.60) | 10.57 (2.94)
  6 Weeks from Baseline: number analyzed (Participants) | 22 | 75 | 73 | 73 | 75 | 71 | 74 | 72
  6 Weeks from Baseline | 10.27 (2.91) | 10.97 (2.99) | 10.62 (3.01) | 10.64 (2.93) | 10.37 (3.09) | 10.90 (2.81) | 10.89 (2.72) | 10.36 (3.19)
  14 Weeks from Baseline: number analyzed (Participants) | 22 | 76 | 78 | 69 | 73 | 74 | 71 | 76
  14 Weeks from Baseline | 9.87 (3.09) | 10.45 (3.28) | 10.45 (3.27) | 9.86 (3.10) | 10.01 (3.28) | 10.32 (3.12) | 10.54 (3.02) | 9.83 (3.33)
Statistical Analysis 1: Comparison: Motivational Interviewing On vs Motivational Interviewing Off vs Personalized Recommendation On vs Personalized Recommendation Off vs Psychoeducation On vs Psychoeducation Off vs Repeated Administration On vs Repeated Administration Off; This analysis explores the time effect of attitudinal changes over the 14 week course of the study, regardless of the combination of components participants were assigned (ie., component turned off or on). Results will help determine whether mean participant attitudes toward change for concerns related to their eating, weight, and/or shape concerns varied based on the time elapsed since engagement with the intervention (ie., do attitudinal changes post-inntervention endure over time?); Test type: Superiority — [test comment as in outcome 2, analysis 2]; p < .001, Linear Mixed Effects Model — We computed both unstandardized (B) and standardized (ß) coefficients to indicate effect sizes. As suggested by Fey et al. (2023), we interpreted absolute ß values below 0.2 as small, between 0.2 and 0.5 as medium, and greater than 0.5 as large; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -.07, Standard Error of Mean .02
Statistical Analysis 2: Comparison: Motivational Interviewing On vs Motivational Interviewing Off; Analyses were conducted to determine the interaction effects of time since intervention and each of the four chatbot components. This analysis explores the interaction effects of time and the motivational interviewing (MI) component on participant attitudes toward change for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = .026, Linear Mixed Effects Model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -0.06, Standard Error of Mean .03
Statistical Analysis 3: Comparison: Personalized Recommendation On vs Personalized Recommendation Off; Analyses were conducted to determine the interaction effects of time since intervention and each of the four chatbot components. This analysis explores the interaction effects of time and the personalized recommendation (PR) component on participant attitudes toward change for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = .465, Linear Mixed Effects Model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = .02, Standard Error of Mean .03
Statistical Analysis 4: Comparison: Psychoeducation On vs Psychoeducation Off; Analyses were conducted to determine the interaction effects of time since intervention and each of the four chatbot components. This analysis explores the interaction effects of time and the psychoeducation (PE) component on participant attitudes toward change for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = .536, Linear Mixed Effects Model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = -.02, Standard Error of Mean .03
Statistical Analysis 5: Comparison: Repeated Administration On vs Repeated Administration Off; Analyses were conducted to determine the interaction effects of time since intervention and each of the four chatbot components. This analysis explores the interaction effects of time and the repeated administration (RA) component on participant attitudes toward change for concerns related to their eating, weight, and/or shape concerns since engagement with the intervention; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = .049, Linear Mixed Effects Model — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 2, analysis 2]; Regression (Beta) Coefficient = .06, Standard Error of Mean .03

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 14-weeks following baseline assessment.
Arm/Group | Repeated Administration | Personalized Recommendation | Motivational Interviewing | Core Modules Only | Motivational Interviewing, Personalized Recommendation, Repeated Administration | Motivational Interviewing, Repeated Administration | Motivational Interviewing, Personalized Recommendation | Personalized Recommendation, Repeated Administration | Psychoeducation | Psychoeducation, Repeated Administration | Psychoeducation, Personalized Recommendation | Psychoeducation, Motivational Interviewing | Psychoeducation, Motivational Interviewing, Personalized Recommendation | Psychoeducation, Personalized Recommendation, Repeated Administration | Psychoeducation, Motivational Interviewing, Repeated Administration | Psychoeducation, Motivational Interviewing, Personalized Recommendation, Repeated Administration
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/14 | 0/13 | 0/13 | 0/14 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13 | 0/13 | 0/13 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/14 | 0/13 | 0/13 | 0/14 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13 | 0/13 | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/11 | 0/14 | 0/13 | 0/13 | 0/14 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13 | 0/13 | 0/13 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04806165/Prot_SAP_ICF_000.pdf